CLINICAL TRIAL: NCT03070834
Title: Retrievable Inferior Vena Cava Filter for Primary Pulmonary Embolism Prophylaxis in At-Risk Trauma Patients: RIPT Feasibility Trial
Brief Title: RIPT Feasibility Trial
Acronym: RIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108169
Record Dates: First submitted 2017-02-17; First posted 2017-03-06 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Embolism; Trauma; Venous Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Wounds and Injuries; Venous Thromboembolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rIVCF (Experimental): Randomized to receive insertion of retrievable inferior vena cava filter until chemical anticoagulation can be safely administered.
  Interventions: Device: Cook 'Celect' retrievable inferior vena cava filter
- Standard Care (No Intervention): Randomized to not receive insertion of retrievable inferior vena cava filter.

INTERVENTIONS:
Device: Cook 'Celect' retrievable inferior vena cava filter — Cook 'Celect' device will be deployed If randomized to rIVCF insertion
  Arms: rIVCF

SUMMARY:
The risk of venous thromboembolism (VTE) is very high in trauma patients, secondary to tissue injury, venous status from immobilization, and thrombophilia. As such, early initiation of VTE prophylaxis is essential in this population. The competing risks of life threatening hemorrhage and VTE need to be considered very carefully. Potential approaches to VTE prophylaxis include pharmacologic means, and mechanical devices. For patients unable to receive pharmacologic VTE prophylaxis, retrievable inferior vena cava filters (rIVCFs) may be placed until low molecular weight heparin (LMWH) can be initiated, as per guidelines such as Eastern Association for the Surgery of Trauma

The investigators propose a feasibility study to determine whether or not our center can insert rIVCFs in at-risk trauma patients expeditiously enough to cause a meaningful reduction in the time they are left unprotected to PE.

DETAILED DESCRIPTION:
The risk of venous thromboembolism (VTE) is very high in trauma patients, secondary to tissue injury, venous status from immobilization, and thrombophilia. As such, early initiation of VTE prophylaxis is essential in this population. The competing risks of life threatening hemorrhage and VTE need to be considered very carefully. Potential approaches to VTE prophylaxis include pharmacologic means, and mechanical devices. For patients unable to receive pharmacologic VTE prophylaxis, retrievable inferior vena cava filters (rIVCFs) may be placed until low molecular weight heparin (LMWH) can be initiated.

The need for mechanical VTE prophylaxis in patients unable to receive pharmacologic therapy is underscored by Geerts and colleagues' prospective study of trauma patients who did not receive anticoagulation. In their study, 58% of their 349 trauma patients sustained deep venous thromboses (DVT). [Geerts et a., 1994] Furthermore, a confirmed or clinically suspected pulmonary embolus (PE) was identified in an additional 5% of patients. Importantly, this study excluded patients who died during the first 5 days of admission. However, the highest risk of VTE occurs in the first 4 days after admission and many advocate early insertion of rIVCF [Owings et al. 1997, O'Malley et al. 1990, Carlin et al. 2002, Haut et al. 2014]. Coincidentally, VTE prophylaxis is often withheld pending repeat neurologic imaging and / or surgical intervention.

Current guidelines on the use of rIVCFs are contradictory. The Eastern Association for the Surgery of Trauma's (EAST) practice management guideline suggests the use of rIVCFs are advisable in the "very-high-risk trauma patients". Such patients are defined as the those who cannot receive anticoagulation because of increased bleeding risk and have sustained injuries preventing mobilization such as: i) severe closed head injury (GCS < 8) ii) incomplete spinal cord injury with paraplegia or quadriplegia iii) complex pelvic fracture with associated long bone fractures iv) multiple long bone fractures [Rogers et al 2002]. Contrasting this, the American College of Chest Physicians sated in their 2012 Guideline, that there is no role for rIVCFs in primary VTE prevention. [Gould et al. 2012]

Reflecting this lack of consensus in guidelines, there is practice variability among major trauma centres. In an American based survey study of 131 Trauma Directors, LMWH was the preferred method for VTE prophylaxis in over half (51%) of the responders, followed by intermittent pneumatic compression devices (IPCD, 42%), Foot pump (8%) Low Dose Heparin (LDH, 7%) and rIVCFs (1%). In patients with contraindications to pharmacologic prophylaxis, the favoured approach for VTE Prophylaxis is IPCD (80%) followed by rIVCF (16%) and foot pump (9%). [Knudson et al. 2004] More work is needed to improve our understanding of the optimal role for rIVCFs, particularly considering recent advances in, and physician experience with rIVCF technology.

One of the most cited concerns with the use of rIVCF in trauma patients is the low reported retrieval rates ranging from 21-35% of patients. [Kirilcuk et al. 2005, Antevil et al. 2006, Karmy-Jones et al., 2007] The need for VTE prophylaxis in trauma patients is usually temporary, and long term filter use is associated with an increased VTE risk, which was demonstrated in the PREPIC-1 trial and the 8-year follow up study examining the use of permanent IVCF in non-trauma patients with DVT for PE prevention [Decousus et al. 1998, PREPIC Study Group, 2005]. Of note, these trials were examining the role of rIVCF in patients for secondary prophylaxis in at risk patients with known VTE disease. The low retrieval rates of rIVCFs that have been reported in the Unites States are not a problem in our Canadian Lead Trauma Centre. We recently demonstrated a 97% retrieval rate in trauma patients surviving to discharge. [Leeper et al. 2015] We advocate a trial of early rIVCF use followed by prompt removal once medical prophylaxis is safe.

There is a paucity of data regarding the use of rIVCFs in the Canadian setting, and our group is currently surveying Canadian trauma directors to improve our understanding of current practice. Despite the current deficiency of evidence, many Level 1 North American Trauma centres use rIVCF for primary VTE prophylaxis in their at risk trauma patients, as per EAST guidelines. In a recent meta-analysis by Haut et al. that reviewed 8 studies, they identified a reduction in PE incidence with rIVCF use, but concluded that further studies are required. [Haut et al. 2014]

The investigators propose a feasibility study to determine whether or not our center can insert rIVCFs in at-risk trauma patients expeditiously enough to cause a meaningful reduction in the time they are left unprotected to PE.

ELIGIBILITY:
Inclusion Criteria:

* consecutive age adult trauma patients who are:

  1. Deemed unable to receive medial VTE prophylaxis within 72 hours post injury based on traumatologists' suspicion of increased bleeding risk, peri-spinal cord bleeding risk, or need for multiple surgical interventions.

     AND
  2. have at-least on of the following high risk VTE injuries as per EAST Guidelines:

     1. severe closed head injury (GCS 8 or less upon presentation)
     2. incomplete spinal cord injury with paraplegia or quadriplegia
     3. complex pelvic fracture with associated long bone fracture(s)
     4. multiple long bone fractures

Exclusion Criteria:

1. Patients not expected to survive for at least 72 hours post trauma
2. Patients with known uncorrectable coagulopathy
3. Patients known to be unable to receive a rIVC filter as part of this trial (for anatomical reasons or standard contraindication for device insertion)
4. Known active venous thromboembolic disease
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Time left unprotected to venous thromboembolism | two weeks post trauma
  time left unprotected to pulmonary embolism two weeks post arrival to hospital defined as: time point from arrival to LHSC to two weeks after, measured in hours where-in patient either has no rIVCF in situ, or has no regular low molecular weight heparin (LMWH) on board. missed doses of LMWH > 2 hours within planned administration time will count toward primary outcome. If LMWH is held for operative intervention, time left held > 24 hours post previous dose will count toward the primary outcome.

SECONDARY OUTCOMES:
Venous Thromboembolism | in hospital (up to one year)
  1. Incidence of symptomatic/clinically impactful pulmonary embolism (as defined by result of computed tomography pulmonary angiogram, autopsy, or ventilation perfusion scan, reported by a radiologist and ordered at the discretion of the MRP on clinical grounds.
Mortality | In Hospital (up to one year)
  in hospital death
Filter Feasibility Outcome: Time to filter insertion | hours to weeks, up to one year
  a) time to filter insertion (defined as time from arrival to London Health Sciences Cente, to time of insertion of rIVCF as documented on the procedure note) b) time to filter removal (defined as time from rIVCF insertion, to removal) c) filter retrieval rate (percentage of patients who receive rIVCF who have rIVCF extraction, will track all patients through follow-up in Trauma Clinic upon discharge if they still have their devices in-situ)
Filter Feasibility Outcome: Time to filter removal | hours to weeks, up to one year
  b) time to filter removal (defined as time from rIVCF insertion, to removal)
Filter Feasibility Outcome: Filter retrieval rate | hours to weeks, up to one year
  c) filter retrieval rate (percentage of patients who receive rIVCF who have rIVCF extraction, will track all patients through follow-up in Trauma Clinic upon discharge if they still have their devices in-situ)
Rates of worsening intracranial bleed | up to 2 weeks
  5) rates of worsening intracranial haemorrhage within patients: Defined as the change in cubic volume of the documented hematoma found in serial computed tomography investigations (if done so as part of routine care)

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Result] Geerts WH, Code KI, Jay RM, Chen E, Szalai JP. A prospective study of venous thromboembolism after major trauma. N Engl J Med. 1994 Dec 15;331(24):1601-6. doi: 10.1056/NEJM199412153312401. PMID 7969340
- [Result] Owings JT, Kraut E, Battistella F, Cornelius JT, O'Malley R. Timing of the occurrence of pulmonary embolism in trauma patients. Arch Surg. 1997 Aug;132(8):862-6; discussion 866-7. doi: 10.1001/archsurg.1997.01430320064010. PMID 9267270
- [Result] O'Malley KF, Ross SE. Pulmonary embolism in major trauma patients. J Trauma. 1990 Jun;30(6):748-50. doi: 10.1097/00005373-199006000-00018. PMID 2352304
- [Result] Carlin AM, Tyburski JG, Wilson RF, Steffes C. Prophylactic and therapeutic inferior vena cava filters to prevent pulmonary emboli in trauma patients. Arch Surg. 2002 May;137(5):521-5; discussion 525-7. doi: 10.1001/archsurg.137.5.521. PMID 11982463
- [Result] Haut ER, Garcia LJ, Shihab HM, Brotman DJ, Stevens KA, Sharma R, Chelladurai Y, Akande TO, Shermock KM, Kebede S, Segal JB, Singh S. The effectiveness of prophylactic inferior vena cava filters in trauma patients: a systematic review and meta-analysis. JAMA Surg. 2014 Feb;149(2):194-202. doi: 10.1001/jamasurg.2013.3970. PMID 24195920
- [Result] Rogers FB, Cipolle MD, Velmahos G, Rozycki G, Luchette FA. Practice management guidelines for the prevention of venous thromboembolism in trauma patients: the EAST practice management guidelines work group. J Trauma. 2002 Jul;53(1):142-64. doi: 10.1097/00005373-200207000-00032. No abstract available. PMID 12131409
- [Result] Gould MK, Garcia DA, Wren SM, Karanicolas PJ, Arcelus JI, Heit JA, Samama CM. Prevention of VTE in nonorthopedic surgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e227S-e277S. doi: 10.1378/chest.11-2297. PMID 22315263
- [Result] Knudson MM, Ikossi DG, Khaw L, Morabito D, Speetzen LS. Thromboembolism after trauma: an analysis of 1602 episodes from the American College of Surgeons National Trauma Data Bank. Ann Surg. 2004 Sep;240(3):490-6; discussion 496-8. doi: 10.1097/01.sla.0000137138.40116.6c. PMID 15319720
- [Result] Kirilcuk NN, Herget EJ, Dicker RA, Spain DA, Hellinger JC, Brundage SI. Are temporary inferior vena cava filters really temporary? Am J Surg. 2005 Dec;190(6):858-63. doi: 10.1016/j.amjsurg.2005.08.009. PMID 16307934
- [Result] Antevil JL, Sise MJ, Sack DI, Sasadeusz KJ, Swanson SM, Rivera L, Lome BR, Weingarten KE, Kaminski SS. Retrievable vena cava filters for preventing pulmonary embolism in trauma patients: a cautionary tale. J Trauma. 2006 Jan;60(1):35-40. doi: 10.1097/01.ta.0000197607.23019.ab. PMID 16456434
- [Result] Karmy-Jones R, Jurkovich GJ, Velmahos GC, Burdick T, Spaniolas K, Todd SR, McNally M, Jacoby RC, Link D, Janczyk RJ, Ivascu FA, McCann M, Obeid F, Hoff WS, McQuay N Jr, Tieu BH, Schreiber MA, Nirula R, Brasel K, Dunn JA, Gambrell D, Huckfeldt R, Harper J, Schaffer KB, Tominaga GT, Vinces FY, Sperling D, Hoyt D, Coimbra R, Rosengart MR, Forsythe R, Cothren C, Moore EE, Haut ER, Hayanga AJ, Hird L, White C, Grossman J, Nagy K, Livaudais W, Wood R, Zengerink I, Kortbeek JB. Practice patterns and outcomes of retrievable vena cava filters in trauma patients: an AAST multicenter study. J Trauma. 2007 Jan;62(1):17-24; discussion 24-5. doi: 10.1097/TA.0b013e31802dd72a. PMID 17215729
- [Result] Decousus H, Leizorovicz A, Parent F, Page Y, Tardy B, Girard P, Laporte S, Faivre R, Charbonnier B, Barral FG, Huet Y, Simonneau G. A clinical trial of vena caval filters in the prevention of pulmonary embolism in patients with proximal deep-vein thrombosis. Prevention du Risque d'Embolie Pulmonaire par Interruption Cave Study Group. N Engl J Med. 1998 Feb 12;338(7):409-15. doi: 10.1056/NEJM199802123380701. PMID 9459643
- [Result] PREPIC Study Group. Eight-year follow-up of patients with permanent vena cava filters in the prevention of pulmonary embolism: the PREPIC (Prevention du Risque d'Embolie Pulmonaire par Interruption Cave) randomized study. Circulation. 2005 Jul 19;112(3):416-22. doi: 10.1161/CIRCULATIONAHA.104.512834. Epub 2005 Jul 11. PMID 16009794
- [Result] Leeper WR, Murphy PB, Vogt KN, Leeper TJ, Kribs SW, Gray DK, Parry NG. Are retrievable vena cava filters placed in trauma patients really retrievable? Eur J Trauma Emerg Surg. 2016 Aug;42(4):459-464. doi: 10.1007/s00068-015-0553-5. Epub 2015 Jul 23. PMID 26201391
- [Derived] Young T, Sriram KB. Vena caval filters for the prevention of pulmonary embolism. Cochrane Database Syst Rev. 2020 Oct 8;10(10):CD006212. doi: 10.1002/14651858.CD006212.pub5. PMID 33027844